CLINICAL TRIAL: NCT06050993
Title: Exploration of Primary Haemostasis in Cirrhotic Patients With T-TAS System and Effects of Platelets Mimicking Nanoparticles
Brief Title: Effects of Platelet Mimicking Nanoparticles in Patients With Cirrhosis
Acronym: HEMCITAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Société Française d'Anesthésie et de Réanimation (Other); CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP230249; 2023 -A00064-41 (Other: IDRCB)
Record Dates: First submitted 2023-07-07; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-07

CONDITIONS: Liver Cirrhosis
Keywords: Hemostatics; Blood Coagulation Disorders; Liver Cirrhosis; Platelet Adhesiveness
MeSH Terms: conditions — Liver Cirrhosis; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 additional citrate tubes (total volume : 9 ml) and 1 Benzylsulfonyl-D-Arg-Pro-4-amidinobenzylamide (BAPA) tube (total volume : 3 ml) will be withdrawn at the same time and in addition of those already withdrawn for the patient's standard of care.
  Plasma aliquots will be done from citrate tubes and frozen. Whole blood tube will be used on the same day of sampling.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cirrhotic patients: Patients known to have a cirrhosis, with an invasive procedure scheduled at the Paul Brousse hospital
  Interventions: Other: Additional blood sampling at the same time and in addition of samplings already done for the patient's standard of care.
- Non-cirrhotic patients: Patients without cirrhosis, with an invasive procedure scheduled at the Paul Brousse hospital
  Interventions: Other: Additional blood sampling at the same time and in addition of samplings already done for the patient's standard of care.

INTERVENTIONS:
Other: Additional blood sampling at the same time and in addition of samplings already done for the patient's standard of care. — During the preoperative procedure scheduled at the Paul Brousse hospital, 3 additional blood tubes (total volume 12 ml) will be withdrawn in addition of samplings already done for the patient's standard of care.

SUMMARY:
Haemostasis of cirrhotic patients is disturbed at different levels: primary haemostasis, coagulation and fibrinolysis, leading to a new haemostatic balance. Thrombocytopenia and thrombopathy are counterbalanced by elevation of Von Willebrand factor (VWF) and diminution of ADAMTS13 activity. Exploration of primary haemostasis is difficult in the laboratory, and non-interpretable in case of thrombocytopenia. Moreover, these tests are not performed under flow conditions. The T-TAS®01 system analyses the total haemostatic capacity in whole blood under shear stress, with chips coated with type 1 collagen. Platelets transfusion performs poorly in cirrhotic patients and is not recommended before invasive procedure. Platelets mimicking nanoparticles (PMNs) have been developed by Pr Sen Gupta (Case Western Reserve University, Cleveland, Ohio (OH), USA). PMNs have been proven to collaborate with platelets and enhance haemostasis in different shear conditions in vitro and in different models of haemorrhage in vivo. The assumption of this study is that the perfusions characteristics of cirrhotic patients in the T-TAS®01 system will be different from those of non-cirrhotic patients, and that platelets mimicking nanoparticles will improve these characteristics.

DETAILED DESCRIPTION:
Hepatic cirrhosis is accompanied by an alteration of the haemostatic balance (primary haemostasis, coagulation, fibrinolysis). With regard to primary haemostasis, thrombocytopenia is usually moderate, due to splenic or hepatic sequestration associated with portal hypertension. Platelet synthesis is also reduced. There are also autoimmune thrombocytopenia due to the presence of anti-platelet autoantibodies. In addition, there is a thrombopathy with functional alterations in platelet adhesion and aggregation. In parallel with these abnormalities in platelet adhesion and aggregation, the quantitative increase in the level of Von Willebrand factor (VWF) preserves the capacity for platelet aggregation, even under conditions of circulating flow, despite the reduction in the intrinsic functional capacity of VWF. This increase can be explained by increased hepatic synthesis, a larger endothelial surface area in the presence of collateral circulation and repeated endothelial aggression by endotoximia during infections, as well as a decrease in clearance due to a decrease in the synthesis of ADAMTS13.

Routine investigation of abnormalities in primary haemostasis is based almost exclusively on platelet counts, as well as plasma VWF and ADAMTS13 assays. Functional platelet tests (PFA®, impedance aggregometry, light transmission aggregation) are more difficult to perform, particularly in the case of thrombocytopenia, and are not performed under circulating flow conditions. The Total Thrombus Formation Analysis System (T-TAS®01) allows analysis of haemostatic capacity in whole blood and flow conditions. Whole blood is deposited in a reservoir and then perfused onto a type I collagen-coated chip (PL chip) at a shear rate of 1500 s-1, mimicking blood flow in small arteries. As the clot forms, the pressure in the perfusion chamber increases until total occlusion occurs. The parameters measured are :

* the time required to achieve a pressure within the perfusion chamber equal to 10 kilopascal (kPa) above the baseline pressure,
* the time required to reach a pressure of 60 kPa above the base pressure in the infusion chamber (occlusion time)
* the area under the curve at 10 min. The perioperative management of cirrhotic patients leads the clinician to ask the question of prophylactic platelet transfusion in the event of thrombocytopenia of less than 30 to 50 G/L. While this threshold value is based on a low level of evidence, platelet transfusion has a poor performance in cirrhotic patients and is not without side effects. Thus, preventive platelet transfusion is not recommended. In the event of bleeding, management should consist of platelet transfusion, combined with fibrinogen and antifibrinolytic administration. Synthetic platelet mimicking particles (SPs) are made of a liposomal membrane, and "decorated" with 3 different peptides: collagen binding peptide (CBP), which binds to fibrillar collagen exposed at the subendothelium, fibrinogen mimetic peptide (FMP), which can bind to the active form of platelet integrin αIIbβ3, and VWF binding peptide (VBP), which is derived from the C2 domain of factor VIII and can bind to the D'-D3 domain of VWF.

Ex vivo, in the absence of endothelial injury, these SPs do not induce platelet aggregation in the absence of agonist but enhance aggregation in the presence of agonist. These SPs do not trigger thrombin formation on their own but in the presence of tissue factor SPs increase thrombin generation and fibrin formation. In perfusion chambers, these nanoparticles allow platelets to adhere to a collagen-coated surface and to aggregate with each other. In vivo, SPs collaborate with platelets to restore effective haemostasis in thrombocytopenic mice undergoing tail-clipping. Their haemostatic efficacy has also been demonstrated in various animal models of traumatic injury, including a mouse model of liver laceration, a porcine model of traumatic arterial haemorrhage, and a rodent model of liver resection.

The assumption of this study is that the characteristics of infusions with the T-TAS®01 system will be altered in cirrhotic patients, reflecting impairment of primary haemostasis, compared to control patients and that platelet-mimicking nanoparticles (PMNs) will correct these alterations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are beneficiaries of a social security scheme or beneficiaries entitled to it
* Patients followed for a cirrhotic pathology at the Paul Brousse hospital and benefiting from a scheduled anaesthesia consultation for a scheduled interventional or surgical procedure
* For non-cirrhotic patients: adult patients who are beneficiaries of a social security scheme or beneficiaries entitled to it, benefiting from a blood test scheduled as part of their usual preoperative care (patients in the hepatology or digestive surgery department operated on at the Paul Brousse hospital)

Exclusion Criteria:

* Patient not wishing to participate in the study
* Patient with a known haemostasis abnormality other than cirrhosis
* Patient on long-term antiplatelet or anticoagulant therapy
* Patient who has taken a non-steroidal anti-inflammatory drug within 5 days prior to the blood test
* Patients with thrombopathy of genetic origin
* Patient on estrogenic therapy
* Patient with cancer under treatment or treated in the last 6 months
* Patient on immunosuppressive or immunomodulatory therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients coming to the Paul Brousse hospital for a scheduled preoperative procedure.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Area under the curve at 10 min of the T-TAS® 01 perfusion in PL chips | One day

SECONDARY OUTCOMES:
Time to reach a pressure of 10 kPa above baseline | One day
Time to reach a pressure of 60 kPa above baseline | One day
Correlations between laboratory results and perfusions' characteristics | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Anaesthesia unit of the Hepatobiliary Center - Paul Brousse Hospital, Villejuif, France

IPD SHARING:
Plan to Share IPD: No